CLINICAL TRIAL: NCT03960931
Title: Interest of Hydrophysiotherapy Care in Parkinson Disease's Non-motor Symptoms
Brief Title: Interest of Hydrophysiotherapy Care in Parkinson Disease's Motor and Non-motor Symptoms
Acronym: THERMAPARK
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: Institut Régional de Médecine Physique et de Réadaptation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2019-A00753-54
Record Dates: First submitted 2019-04-12; First posted 2019-05-23 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Interest of Hydrophysiotherapy Care in Parkinson Disease's Non-motor Symptoms
Keywords: Parkinson's disease; Non motor signs; Postural control; Gait; Hydrophysiotherapy
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Aquatic rehabilitation (Experimental)
  Interventions: Other: Aquatic rehabilitation
- Land based physical activities (Experimental)
  Interventions: Other: Land based physical activities
- Conventional rehabilitation (Other)
  Interventions: Other: Conventional rehabilitation

INTERVENTIONS:
Other: Aquatic rehabilitation — Rehabilitation sessions using hydrophysiotherapy will occur in a pool of Grand Nancy Thermal, three times per week during 4 weeks, and each will last 45 min. They will begin with 10 min of warm-up, then 30 min of walking. Sessions will end cool-down during 5 min, which will be a reduction of intensity every 30 sec. Rehabilitation will be carried out by physiotherapist chosen for the study.
  Other Names: Hydrophysiotherapy
  Arms: Aquatic rehabilitation
Other: Land based physical activities — Rehabilitation sessions on treadmill will occur at Physical Medicine and Rehabilitation Regional Institute (IRR), on the University Hospital's site, three times per week during 4 weeks, and each will last 45 min. They will begin with 10 min of warm-up, then 30 min of walking, where intensity of effort can be modulated by speed and inclination of treadmill. Sessions will end cool-down during 5 min, which will be a reduction of intensity every 30 sec. Rehabilitation will be carried out by physiotherapist chosen for the study.
  Arms: Land based physical activities
Other: Conventional rehabilitation — Conventional rehabilitation sessions will occur in private practices in which patients receive their habitual care (same physiotherapist). This care will be guided by prescription delivered by the neurologist. This prescription suggests to work on active and passive upper and lower limb stretching, on hip and shoulder dissociation, and balance control management on unstable ground.
  Arms: Conventional rehabilitation

SUMMARY:
Parkinson Disease (PD) is a neurodegenerative disorder who begin around 55 years old, characterized by brain's backmatter's dopamine neuron destruction, involved in motor control. Diagnosis is made with presence of 3 of 4 disease's cardinal sign: bradykinesia, rigidity, resting tremor, walking troubles. Treatments enhance patient's quality of life, but do not allow to stop disease's evolution, who is specific depending on a lot of factors. For some years, PD's non motor symptoms (NMS) - in particular pain, anxiety, depression, sleep disorders - have been highlighted and turn out to impair sometimes quality of life even though motor symptoms are controlled. This project's main aim is to evaluate if aquatic environment's care lead to an advantage on PD's NMS, symptoms currently underestimated, insufficiently in care and having a harmful influence on quality of life. Collaboration of the University Hospital (Neurology Dpt), the Physical Medicine and Rehabilitation Regional Institute, Grand Nancy Thermal, and France Parkinson Association, will allow in this way to offer on PD's NMS, postural control impairments, and walking troubles an alternative or further non-pharmacological therapy.

ELIGIBILITY:
Inclusion Criteria, patient:

* having get a complete information on study's organization and having given written informed consent,
* affiliated to a social security system,
* suffering from Parkinson's disease (stage 2 or 3 of Hoehn and Yahr),
* with motor fluctuation lower than 25% of awaked time,
* with dyskinesia lower than 25% of awaked time (according to MDS-UPDRS scale),
* with stable pharmacological treatment during the 30 days before study,
* already benefiting of a physiotherapy.

Exclusion Criteria, patients:

* receiving treatment by apomorphine or Duodopa pump,
* benefiting of brain stimulation,
* taking occasionally benzodiazepine,
* with dementia (MDS-UPDRS 1.1 score > 3),
* having had a sprain on a lower limb joint 3 months or less before the beginning of study,
* having head trauma consequences,
* having vertebrae pain,
* with freezing,
* having skin trouble leading to a contraindication of aquatic activities,
* concerned by L. 1121-5, L. 1121-7 and L 1121-8 articles of French public health code.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2019-07-01 (Estimated); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-11-30 (Estimated)

PRIMARY OUTCOMES:
Change of score on Parkinson's Disease Questionnaire 39 (PDQ 39) after reeducation | Day 1, day 28 (+7)
  Total score to PDQ 39 (between 0 and 156, a lower score being a better outcome), which evaluates quality of life, before and after reeducation

SECONDARY OUTCOMES:
Persistence of change of score on PDQ 39 after reeducation | Day 28(+7), day 56 (+/-7)
  Total score to Parkinson Disease Questionnaire 39 (between 0 and 156, a lower score being a better outcome), which evaluates quality of life, before and after reeducation.
PDQ 39 sub-scores | Day 1, day 28 (+7), day 56 (+/-7)
  Sub-score for each of the 8 fields composing PDQ 39: mobility, activities of daily living, emotional well-being, stigma, social support, cognition, communication and bodily discomfort
Non-Motors Signs (NMS) Questionnaire score | Day 1, day 28 (+7), day 56 (+/-7)
  Questionnaire score for NMS (non motor signs) in its globality.
Parkinson Anxiety Scale (PAS) score | Day 1, day 28 (+7), day 56 (+/-7)
  Parkinson's Anxiety Scale, evaluating anxiety (between 0 and 30, a lower score being a better outcome).
Parkinson's Disease specific Pain score | Day 1, day 28 (+7), day 56 (+/-7)
  King's Parkinson's Disease Pain Scale (KPPS, between 0 and 168, a lower score being a better outcome)
Global Pain score | Day 1, day 28 (+7), day 56 (+/-7)
  Visual Analogic Scale (VAS) (between 0 and 10, a lower score being a better score)
Mean Equilibrium path length | Day 1, day 28 (+7), day 56 (+/-7)
  Corresponding to the mean path length travelled by displacement of the Centre of Foot Pressure in four conditions (eyes open or closed, firm or foamed support).
Mean Equilibrium ellipse area | Day 1, day 28 (+7), day 56 (+/-7)
  Corresponding to the mean ellipse area covered by displacement of the Centre of Foot Pressure in four conditions (eyes open or closed, firm or foamed support)
Ratio of sensory inputs. | Day 1, day 28 (+7), day 56 (+/-7)
  Ratio of sensory inputs in postural control (somatosensory, visual and vestibular ratios).
Entropy | Day 1, day 28 (+7), day 56 (+/-7)
  Entropy mathematically evaluates the displacements regularity of the Center of Foot Pressure (CoP). If the CoP displacements are regular (lower entropy), intentionally processes are more implicated in postural control regulation. If the CoP displacements are not regular (higher entropy), automatic processes are more implicated in postural control regulation. Entropy comparison between a single and a dual task is analyzed.
Time for Time Up and Go (TUG) | Day 1, day 28 (+7), day 56 (+/-7)
  Timed Up and Go
Distance of walking | Day 1, day 28 (+7), day 56 (+/-7)
  Distance walked during the 6 min walk test
Walking velocity | Day 1, day 28 (+7), day 56 (+/-7)
  Mean velocity during the 6 min walk test.
Step high | Day 1, day 28 (+7), day 56 (+/-7)
  Mean step high during the 6 min walk test.
Step length | Day 1, day 28 (+7), day 56 (+/-7)
  Mean step length during the 6 min walk test.
Step width | Day 1, day 28 (+7), day 56 (+/-7)
  Mean step width during the 6 min walk test.
Subjective effort | Day 1, day 28 (+7), day 56 (+/-7)
  Ratio of Perceived Exertion (RPE) score, evaluated by Borg Scale (according to the 6 min walk test). Score is between 6 and 20, 6 being a better outcome.

REFERENCES:
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD013856. doi: 10.1002/14651858.CD013856.pub3. PMID 38588457
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886